CLINICAL TRIAL: NCT02079636
Title: A Phase 1b Study of LY2835219 in Combination With Multiple Single Agent Options for Patients With Stage IV NSCLC
Brief Title: A Study of Abemaciclib (LY2835219) in Combination With Another Anti-cancer Drug in Participants With Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15266; I3Y-MC-JPBJ (Other: Eli Lilly and Company); 2013-004648-41 (EudraCT Number); KEYNOTE-238 (Other: Merck)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2019-11-15

CONDITIONS: Carcinoma, Non-small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abemaciclib; Pemetrexed; Gemcitabine; Ramucirumab; LY3023414; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Abemaciclib + Pemetrexed (Experimental): 150 milligram (mg) or 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 500 milligrams/square meter (mg/m^2) pemetrexed given intravenously (IV) over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Pemetrexed
- Abemaciclib + Gemcitabine (Experimental): 150 mg or 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 milligram/square meter (mg/m^2) gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Gemcitabine
- Abemaciclib + Ramucirumab (Experimental): 150 mg or 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 or 8 to 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Ramucirumab
- Abemaciclib + LY3023414 (Experimental): 100 mg or 150 mg or 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100, 150, or 200 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: LY3023414
- Abemaciclib + Pembrolizumab (Experimental): 100 mg or 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 200 mg pembrolizumab given intravenously over approximately 30 minutes on day 1 of a 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
  Interventions: Drug: Abemaciclib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Pemetrexed — Administered IV
  Other Names: Alimta
  Arms: Abemaciclib + Pemetrexed
Drug: Gemcitabine — Administered IV
  Other Names: Gemzar
  Arms: Abemaciclib + Gemcitabine
Drug: Ramucirumab — Administered IV
  Other Names: Cyramza
  Arms: Abemaciclib + Ramucirumab
Drug: LY3023414 — Administered orally
  Arms: Abemaciclib + LY3023414
Drug: Pembrolizumab — Administered IV
  Other Names: Keytruda
  Arms: Abemaciclib + Pembrolizumab

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of abemaciclib in combination with another anti-cancer drug in participants with NSCLC that is advanced or has spread to other parts of the body (stage IV). The study will also investigate how the body processes the combination treatment and how the study drug affects the body. The study will also collect disease-related symptoms and participant-reported pain related to NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* For all Parts: The participant must have stage IV non-small cell lung cancer (NSCLC).
* For Part A (abemaciclib + pemetrexed): Non-squamous subtypes only. The participant must have received at least one but no more than three prior therapies for advanced/metastatic NSCLC.
* For Part B (abemaciclib + gemcitabine): Any subtype. The participant must have received at least one but not more than three prior therapies for advanced/metastatic NSCLC.
* For Part C (abemaciclib + ramucirumab): Any subtype. The participant must have received at least two but not more than three prior therapies for advanced/metastatic NSCLC.
* For Part D (abemaciclib + LY3023414): Any subtype. The participant must have received at least two, but not more than three prior therapies for advanced/metastatic NSCLC. The participant must not have received prior treatment with any phosphoinositide 3-kinase (PI3K) or mammalian target of rapamycin (mTOR) inhibitor.
* For Part E (abemaciclib + pembrolizumab): Any subtype. The participant must have received at least one but no more than three prior therapies for advanced/metastatic NSCLC.
* Have either measureable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
* Have adequate organ function including:

  * Hematologic: Absolute neutrophil count (ANC) 1.5 x 109/liter (L), platelets 100 x 109/L, and hemoglobin 8 gram/deciliter (g/dL).
  * Hepatic: Bilirubin 1.5 times upper limits of normal (ULN), alanine aminotransferase (ALT) and aspartate transaminase (AST) 3.0 times ULN. For participants with tumor involvement of the liver, AST and ALT equaling ≤5.0 times ULN are acceptable. Alkaline phosphatase ≤5.0 times ULN for participants with tumor involvement of the bone is acceptable.
  * Renal: Serum creatinine 1.5 times ULN.
* Have a performance status ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy (treatment related toxicity resolved to baseline) except for residual alopecia.
* Male and female participants of reproductive potential must agree to use medically approved contraceptive precautions during the trial and 3 to 4 months (as appropriate) following last dose of study drug.
* Have an estimated life expectancy of ≥12 weeks.
* Are able to swallow oral medications.

Exclusion Criteria:

* Have a personal history of any of the following conditions: presyncope or syncope of either unexplained or cardiovascular etiology, ventricular arrhythmia (including but not limited to ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest. Exception: Participants with controlled atrial fibrillation for >30 days prior to study treatment are eligible.
* Parts A, B, D and E: Have central nervous system (CNS) metastasis with development of associated neurological changes 14 days prior to receiving study drug.
* Have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix or breast), unless in complete remission with no therapy for a minimum of 3 years.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 3 to 4 months after the last dose of trial treatment (as appropriate).
* Have active bacterial, fungal, and/or known viral infection (for example, human immunodeficiency virus [HIV] antibodies, hepatitis B surface antigen [HBSAg], or hepatitis C antibodies). Screening is not required for enrollment.
* Parts A, B, C, and E: Have QTc interval of > 470 millisecond (msec) on screening electrocardiogram (ECG). Part D participants have QTc interval of >450msec on screening ECG.

Additional Exclusion Criteria For Part C

* History or evidence of cardiovascular risk including any of the following:

  * History of acute coronary syndromes (including myocardial infarction and angina), coronary angioplasty, or stenting within 6 months prior to enrollment.
  * History or evidence of current ≥Class II congestive heart failure as defined by New York Heart Association.
  * Treatment refractory hypertension defined as a blood pressure of systolic >140 millimeter of mercury (mmHg) and/or diastolic >90 mmHg which cannot be controlled by antihypertensive therapy.
  * Participants with intracardiac defibrillators.
* History or evidence of CNS disease. Radiographic screening of all participants without history of CNS metastasis is required.
* Radiographically documented evidence of major vessel invasion or encasement by cancer.
* Uncontrolled thromboembolic or hemorrhagic disorders.
* Participants receiving daily treatment with aspirin >325mg/day or other known inhibitors of platelet function.
* History of gross hemoptysis within 2 months of study entry.
* Evidence of nonhealing wounds, ulcers, or bone fractures within 28 days prior to study entry.
* Undergone major surgery within 28 days prior to first dose of study drug or have subcutaneous venous access device placement within 7 days prior to first dose.

Additional Exclusion Criteria For Part D

* Have insulin-dependent diabetes mellitus or a history of gestational diabetes mellitus.
* Participants with a type 2 diabetes mellitus are eligible if adequate control of blood glucose level is obtained by oral anti-diabetic agents as documented by hemoglobin A1c (HbA1c) <7%.
* History or evidence of cardiovascular risk including any of the following -- History of acute coronary syndromes (including myocardial infarction and angina), coronary angioplasty, or stenting within 6 months prior to enrollment.

Additional Exclusion Criteria for Part E

* Received prior monoclonal antibody (mAb) within 4 weeks prior to study.
* Has active autoimmune disease that has required treatment in the past 2 years.
* Has history of interstitial lung disease or pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- United States (8):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - UCLA Department of Medicine-Hematology/Oncology, Los Angeles, California
  - University of California, Davis - Health Systems, Sacramento, California
  - Indiana Cancer Pavilion, Indianapolis, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Carolinas Medical Center, Charlotte, North Carolina
  - The West Clinic, Germantown, Tennessee
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Majadahonda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

REFERENCES:
- [Derived] Kim ES, Kelly K, Paz-Ares LG, Garrido P, Jalal S, Mahadevan D, Gutierrez M, Provencio M, Schaefer E, Shaheen M, Johnston EL, Turner PK, Kambhampati SRP, Beckmann R, Hossain A, John WJ, Goldman JW. Abemaciclib in Combination with Single-Agent Options in Patients with Stage IV Non-Small Cell Lung Cancer: A Phase Ib Study. Clin Cancer Res. 2018 Nov 15;24(22):5543-5551. doi: 10.1158/1078-0432.CCR-18-0651. Epub 2018 Aug 6. PMID 30082474
- [Derived] Gelbert LM, Cai S, Lin X, Sanchez-Martinez C, Del Prado M, Lallena MJ, Torres R, Ajamie RT, Wishart GN, Flack RS, Neubauer BL, Young J, Chan EM, Iversen P, Cronier D, Kreklau E, de Dios A. Preclinical characterization of the CDK4/6 inhibitor LY2835219: in-vivo cell cycle-dependent/independent anti-tumor activities alone/in combination with gemcitabine. Invest New Drugs. 2014 Oct;32(5):825-37. doi: 10.1007/s10637-014-0120-7. Epub 2014 Jun 13. PMID 24919854
- See also: Click here for more information about this study: A Study of Abemaciclib (LY2835219) in Combination With Another Anti-cancer Drug in Participants With Stage IV Non-small Cell Lung Cancer (NSCLC) — https://www.lillytrialguide.com/en-US/studies/non-small-cell-lung-cancer/JPBJ#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who had cycle 1 and had received greater than or equal to (>=) 75% of Abemaciclib drug in cycle 1.
Groups:
- Part A: 150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed: 150 mg abemaciclib given orally every 12 hours (Q12H) on Days 1 through 21 of a 21-day cycle in combination with 500 milligrams/square meter (mg/m^2) pemetrexed given intravenously (IV) over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 500 mg/m^2 pemetrexed given intravenously (IV) over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 mg/m^2 gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 mg/m^2 gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10mg/kg Ramucirumab Day 1: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 8 mg/kg ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 mg/kg ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 100 mg Abemaciclib + 100 mg LY3023414: 100 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 150 mg Abemaciclib + 100 mg LY3023414: 150 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 150 mg Abemaciclib + 150 mg LY3023414: 150 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 150 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 200 mg Abemaciclib + 150 mg LY3023414: 200 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 150 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 150 mg Abemaciclib + 200 mg LY3023414: 150 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 200 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab: 100 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 200 mg pembrolizumab given intravenously over approximately 30 minutes on day 1 of a 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 200 mg pembrolizumab given intravenously over approximately 30 minutes on day 1 of a 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Part A: 150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C: 150 mg Abemaciclib + 10mg/kg Ramucirumab Day 1 | Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1 | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 150 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
Started | 8 | 15 | 3 | 21 | 4 | 19 | 12 | 4 | 3 | 9 | 10 | 6 | 8 | 3 | 17
Received at Least One Dose of Study Drug | 8 | 15 | 3 | 21 | 4 | 19 | 12 | 4 | 3 | 9 | 10 | 6 | 8 | 3 | 17
Completed | 5 | 13 | 3 | 9 | 2 | 13 | 11 | 3 | 3 | 6 | 8 | 4 | 5 | 3 | 12
Not Completed | 3 | 2 | 0 | 12 | 2 | 6 | 1 | 1 | 0 | 3 | 2 | 2 | 3 | 0 | 5
Not completed — Death | 2 | 1 | 0 | 5 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug in Part A, B, C, D and E.
Groups:
- Part A:150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 500 milligrams/square meter (mg/m^2) pemetrexed given intravenously (IV) over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C:150 mg Abemaciclib+10mg/kg Ramucirumab Day1: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 mg/kg ramucirumab given intravenously over approximately 60 minutes on on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Total: Total of all reporting groups
Arm/Group | Part A:150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C:150 mg Abemaciclib+10mg/kg Ramucirumab Day1 | Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1 | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 150 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab | Total
Number analyzed (Participants) | 8 | 15 | 3 | 21 | 4 | 19 | 12 | 4 | 3 | 9 | 10 | 6 | 8 | 3 | 17 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.88 (7.61) | 62.53 (11.19) | 55.00 (8.66) | 63.14 (10.07) | 61.25 (14.24) | 66.11 (9.31) | 63.75 (6.77) | 67.75 (4.92) | 67.00 (9.54) | 57.56 (8.26) | 64.00 (8.41) | 65.50 (7.48) | 60.38 (10.20) | 67.33 (3.51) | 59.76 (9.94) | 62.89 (9.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 0 | 11 | 2 | 10 | 4 | 0 | 1 | 5 | 3 | 2 | 5 | 1 | 10 | 63
  Male | 4 | 10 | 3 | 10 | 2 | 9 | 8 | 4 | 2 | 4 | 7 | 4 | 3 | 2 | 7 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 7
  Not Hispanic or Latino | 8 | 13 | 2 | 20 | 4 | 17 | 11 | 4 | 3 | 9 | 10 | 5 | 7 | 3 | 17 | 133
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 5
  White | 8 | 13 | 3 | 16 | 4 | 18 | 12 | 4 | 2 | 7 | 10 | 5 | 7 | 3 | 16 | 128
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 8 | 2 | 16 | 4 | 15 | 6 | 1 | 3 | 9 | 10 | 6 | 8 | 0 | 3 | 97
  Spain | 2 | 7 | 1 | 5 | 0 | 4 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 3 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT) or DLT-equivalent in Part A, B, C, D and E
Description: A DLT defined as adverse event(AE) occurring between Day 1 and Day 21 of Cycle 1 that was considered at least possibly related to either abemaciclib or the combination therapy and fulfilled a criteria selected (using the National Cancer Institute Common Terminology Criteria for Adverse Events,version 4.0 [NCI-CTCAE v 4.0] [NCI 2009]):Grade(Gr)≥3 nonhematological toxicity,Gr4 thrombocytopenia lasting at least 5 days and/or complicated with bleeding,Gr≥3 febrile neutropenia(ntr) and for Part D participants (pts): Gr3 hyperglycemia (fasting) of <5 days, Gr3 hypertriglyceridemia or hyperlipidemia without optimal treatment.A DLT-equivalent defined as AE that would have met the criteria for DLT if it had occurred during Cycle 1 for pts enrolled in dose-escalation phase,but that occurs between 1)Day 1 and Day 21 of Cycle 2 and beyond for a participant enrolled in dose-escalation phase 2) at any time for a participant in dose-expansion phase.
Time Frame: Baseline through study completion (Up To 15 Months)
Population: All randomized participants who received at least one dose of study drug in Part A, B, C, D and E.
Measure: Count of Participants; unit: Participants
Groups:
- Part C:150 mg Abemaciclib+10 mg/kg Ramucirumab Day 1: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day 1: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A:150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C:150 mg Abemaciclib+10 mg/kg Ramucirumab Day 1 | Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day 1 | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 150 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
Number analyzed (Participants) | 8 | 15 | 3 | 21 | 4 | 19 | 12 | 4 | 3 | 9 | 10 | 6 | 8 | 3 | 17
Participants | 1 | 4 | 0 | 5 | 1 | 4 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 0 | 0

2. Secondary Outcome: Number of Participants Achieving Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR]) in Part A, B, C, D and E
Description: ORR is the best response of CR or PR as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of not-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants with at least 1 measurable lesion, multiplied by 100.
Time Frame: Baseline through study completion (Up To 15 Months)
Population: All randomized participants who received at least one dose of study drug in Part A, B, C, D and E.
Measure: Count of Participants; unit: Participants
Groups:
- Part C:150 mg Abemaciclib+10mg/kg Ramucirumab Day1: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 or 8 to 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day 1: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 8 mg/kg ramucirumab given intravenously over approximately 60 minutes on Day 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A:150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C:150 mg Abemaciclib+10mg/kg Ramucirumab Day1 | Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day 1 | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 150 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
Number analyzed (Participants) | 8 | 15 | 3 | 21 | 4 | 19 | 12 | 4 | 3 | 9 | 10 | 6 | 8 | 3 | 17
Participants | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2

3. Secondary Outcome: Progression Free Survival Time in Part A, B, C, D and E
Description: Progression free survival (PFS) defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date. PFS time was summarized using Kaplan-Meier estimates.
Time Frame: Date of first dose until first documented progression or death (Up To 15 Months)
Population: All randomized participants in Part A, B, C, D and E. Censored participants: Part A= 13, Part B = 7, Part C = 17, Part D = 19, Part E = 10.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Part A:Abemaciclib + 500 mg/m^2 Pemetrexed: 150/200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 500 milligrams/square meter (mg/m^2) pemetrexed given intravenously (IV) over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part B: Abemaciclib + 1250 mg/m^2 Gemcitabine: 150/200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 mg/m^2 gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C:Abemaciclib+ 8/10mg/kg Ramucirumab Day1/8: 150 /200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 8 mg/kg /10 mg/kg ramucirumab / given intravenously over approximately 60 minutes on Day 1 or 8 to 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: Abemaciclib + 100 mg/150 mg/ 200 mg LY3023414: 100 mg/ 150 mg / 200 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100 mg / 150 mg/ 200 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part E: 100 mg/150 mg Abemaciclib + 200 mg Pembrolizumab: 100 mg / 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 200 mg pembrolizumab given intravenously over approximately 30 minutes on day 1 of a 21 day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A:Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C:Abemaciclib+ 8/10mg/kg Ramucirumab Day1/8 | Part D: Abemaciclib + 100 mg/150 mg/ 200 mg LY3023414 | Part E: 100 mg/150 mg Abemaciclib + 200 mg Pembrolizumab
Number analyzed (Participants) | 23 | 24 | 39 | 36 | 20
Months | 5.55 [1.81 to 22.47] | 1.58 [1.18 to 2.46] | 4.83 [1.61 to 7.16] | 1.87 [1.41 to 5.32] | 4.11 [3.02 to NA] — The upper limit of the 95% confidence Interval (CI) was not calculated due to the high censoring rate.

4. Secondary Outcome: Change From Baseline in MD Anderson Symptom Inventory Scale-Lung Cancer (MDASI-LC) in Part A, B, C, D and E
Description: The MDASI-LC is a self-reported lung cancer instrument included 22 items covered by one of the following dimensions: Mean core symptom severity (Core items 1-13: pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, remembering things, lack of appetite, drowsy, dry mouth, sad, vomiting, numbness/tingling), Lung cancer symptoms (3 items: coughing, constipation, sore throat), Mean symptom severity (13 core items plus 3 lung items) and Interference with mood or functional status (6 items: general activity, mood, work, relations with other people, walking, enjoyment of life). The mean of all symptom subscale items was calculated where 0 equals "not present" and 10 equals "as bad as you can imagine." A change from baseline with negative values indicate improvement, positive values indicate worsening.
Time Frame: Baseline, through study completion (Up To 15 Months)
Population: All randomized participants for cycles which at least 25% of participants in each arm have a score. MDASI-LC population included all randomized participants who completed at least 1 baseline assessment followed by at least 1 MDASI-LC result in Part A, B, C, D and E.
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Groups:
- Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 or 8 to 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 8 mg/kg ramucirumab given intravenously over approximately 60 minutes on Day 1 or 8 to 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 mg/kg ramucirumab given intravenously over approximately 60 minutes on Day 1 or 8 to 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A:150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C:150 mg Abemaciclib+10mg/kg Ramucirumab Day1 | Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1 | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 150 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
Number analyzed (Participants) | 8 | 15 | 2 | 21 | 4 | 19 | 12 | 4 | 3 | 9 | 10 | 6 | 8 | 3 | 17
units on a scale
  Mean core symptom severity: number analyzed (Participants) | 6 | 12 | 1 | 14 | 2 | 12 | 9 | 2 | 3 | 5 | 7 | 3 | 4 | 3 | 13
  Mean core symptom severity | -0.16 [-1.46 to 0.31] | 0.89 [-0.96 to 2.24] | -0.54 [-0.54 to -0.54] | -0.08 [-1.54 to 1.08] | -0.35 [-2.47 to 1.77] | 0.61 [-1.04 to 2.70] | -0.64 [-1.54 to 1.23] | -1.39 [-2.31 to -0.46] | 0.61 [-1.85 to 2.15] | 1.89 [1.00 to 3.85] | 1.60 [-1.15 to 2.77] | -0.80 [-2.93 to 0.38] | 0.28 [-1.62 to 2.18] | 0.91 [0.19 to 1.93] | 0.88 [0.47 to 2.08]
  Mean symptom severity: number analyzed (Participants) | 6 | 12 | 1 | 14 | 2 | 12 | 9 | 2 | 3 | 5 | 7 | 3 | 4 | 3 | 13
  Mean symptom severity | -0.05 [-1.43 to 0.68] | 0.83 [-0.86 to 1.82] | -0.44 [-0.44 to -0.44] | -0.03 [-1.44 to 1.19] | -0.41 [-2.31 to 1.50] | 0.72 [-0.88 to 2.41] | -0.61 [-1.25 to 1.06] | -1.01 [-2.13 to 0.12] | 0.64 [-1.63 to 1.94] | 1.86 [1.50 to 3.62] | 1.60 [-0.94 to 2.88] | -0.73 [-2.82 to 0.37] | 0.19 [-1.35 to 1.73] | 0.99 [0.59 to 1.69] | 0.75 [0.56 to 1.94]
  Mean lung cancer symptom: number analyzed (Participants) | 6 | 12 | 1 | 12 | 2 | 13 | 9 | 2 | 3 | 5 | 7 | 3 | 4 | 3 | 13
  Mean lung cancer symptom | 1.22 [-1.00 to 3.33] | 0.71 [-1.00 to 1.00] | 1.67 [1.67 to 1.67] | 0.19 [-1.00 to 1.00] | -0.67 [-1.67 to 0.33] | 1.13 [-1.00 to 2.00] | -0.78 [-3.00 to 0.67] | 3.01 [2.67 to 3.34] | 0.78 [-0.67 to 2.00] | 1.40 [-0.34 to 2.66] | 2.19 [0.67 to 3.33] | -0.44 [-2.33 to 1.34] | 0.67 [-1.00 to 2.34] | 1.67 [0.67 to 2.33] | 0.23 [-1.00 to 1.67]
  Mean interference severity: number analyzed (Participants) | 6 | 12 | 1 | 12 | 2 | 13 | 9 | 2 | 3 | 5 | 7 | 3 | 4 | 3 | 13
  Mean interference severity | 2.32 [1.50 to 4.20] | 0.49 [-3.00 to 3.59] | 0.00 [0.00 to 0.00] | 0.95 [-0.51 to 4.76] | -1.33 [-3.83 to 1.17] | 0.15 [-3.00 to 3.16] | -1.00 [-5.16 to 1.33] | -3.08 [-4.50 to -1.66] | 0.72 [-1.17 to 3.50] | 1.47 [0.17 to 1.67] | 1.81 [-0.83 to 5.17] | -0.22 [-3.17 to 2.17] | -0.38 [-4.25 to 3.50] | 1.44 [0.33 to 2.83] | 1.00 [-1.67 to 2.84]

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib on Day 1 and at Steady State (Cycle 2 Day 1) in Part A , B, C, D and E
Description: Cmax of Abemaciclib on day 1 and at steady State (Cycle 2 Day 1) Part A , B, C, D and E was evaluated.
Time Frame: Cycle 1 Day 1 (C1D1) pre-dose and 1, 2, 4, 6, 8, 10 h post-dose; Cycle 2 Day 1 (C2D1) pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part A , B, C, D and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 500 mg/m^2 pemetrexed given IV over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 8 mg/kg or 10 mg/kg Ramucirumab: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1, or 8 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8, or 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day 1: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 150 mg Abemaciclib + 100 or 150 or 200 mg LY3023414: 150 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100 or 150 or 200 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C: 150 mg Abemaciclib + 8 mg/kg or 10 mg/kg Ramucirumab | Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day 1 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 or 150 or 200 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
Number analyzed (Participants) | 8 | 15 | 3 | 20 | 20 | 19 | 3 | 27 | 6 | 3 | 17
nanograms per milliliter (ng/mL)
  Day 1 | 114 (67.4) | 212 (79.8) | 80.6 (14.7) | 201 (71.7) | 140 (95.7) | 195 (85.8) | 86.2 (91.1) | 159 (74.1) | 225 (103) | 125 (57.2) | 114 (68.8)
  Steady State: number analyzed (Participants) | 2 | 8 | 2 | 3 | 11 | 6 | 3 | 10 | 0 | 3 | 10
  Steady State | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 146 ng/mL and 183 ng/mL. | 509 (40.5) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 308 ng/mL and 606 ng/mL. | 417 (77.7) | 322 (112) | 228 (152) | 227 (85.1) | 305 (55.8) |  | 270 (47.7) | 240 (87.5)

6. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Pemetrexed at Steady State in Part A
Description: Cmax of pemetrexed at steady state in Part A was evaluated.
Time Frame: C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed
Number analyzed (Participants) | 7 | 12
microgram per milliliter (μg/mL) | 98.1 (29) | 93.5 (30)

7. Secondary Outcome: PK: Dose-normalized Maximum Concentration (Cmax) of Active Gemcitabine Metabolite: 2',2'-Difluorodeoxyuridine (dFdU) on Day 1 and at Steady State (Cycle 2 Day 1) in Part B
Description: Cmax of active gemcitabine metabolite (dFdU) on day 1 and at steady state (Cycle 2 Day 1) dose-normalized to 1250 mg/m^2 in Part B was evaluated.
Time Frame: C1D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose; C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Part B: 200 mg or MTD Abemaciclib + 1250 mg/m^2 Gemcitabine: 200 mg abemaciclib or maximum tolerated dose (MTD) under the combination treatment abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 mg/m^2 gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg or MTD Abemaciclib + 1250 mg/m^2 Gemcitabine
Number analyzed (Participants) | 3 | 4 | 16
nanogram per milliliter (ng/mL)
  Day 1 | 35600 (14) | 49600 (12) | 41900 (21)
  Steady State: number analyzed (Participants) | 2 | 3 | 8
  Steady State | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of Cmax = 33414 ng/mL, 49416 ng/mL. | 38700 (18) | 35800 (17)

8. Secondary Outcome: PK: Maximum Concentration (Cmax) of Ramucirumab at 1 Hour Post-End-of-Infusion in Part C
Description: Cmax of ramucirumab at 1 hour post-end-of-Infusion in Part C was evaluated.
Time Frame: C1D1 and C2D1: 1 hour post-end-of-infusion
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part C.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Groups:
- Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 8 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Day 1: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 milligram/kilogram (mg/kg) ramucirumab given intravenously over approximately 60 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Day 1 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1
Number analyzed (Participants) | 12 | 4 | 4 | 18
microgram per milliliter (μg/mL)
  C1D1 | 174 (19.6) | 226 (10.0) | 193 (27.0) | 221 (30.6)
  C2D1: number analyzed (Participants) | 9 | 2 | 1 | 7
  C2D1 | 221 (15.0) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of Cmax = 283 μg/mL and 264 μg/mL. | NA (NA) — Data reported as individual values when participants analyzed (n) were less than 3. Individual value of Cmax = 158 μg/mL. | 226 (32.3)

9. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3023414 in Part D
Description: Cmax of LY3023414 in Part D was evaluated.
Time Frame: C1D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose; C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part D: 100 or 150 mg Abemaciclib + 100 mg LY3023414: 100 or 150 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part D: 150 or 200 mg Abemaciclib + 150 mg LY3023414: 150 or 200 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 150 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part D: 100 or 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 or 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414
Number analyzed (Participants) | 12 | 15 | 8
nanograms per milliliter (ng/mL)
  Day 1 | 298 (104) | 454 (81) | 578 (119)
  Steady State: number analyzed (Participants) | 12 | 4 | 1
  Steady State | 438 (63) | 491 (52) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of Cmax = 165 ng/mL.

10. Secondary Outcome: PK: Area Under the Concentration Curve (AUC) of Abemaciclib in Part A, B, C, D and E
Description: Area under the concentration time curve from zero to 8 hours AUC(0-8h) of abemaciclib in Part A, B, C, D and E was evaluated.
Time Frame: C1D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose; C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part A, B, C, D and E.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL (ng*h/mL)
Arm/Group | Part A:150 Milligram(mg) Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C: 150 mg Abemaciclib + 8 mg/kg or 10 mg/kg Ramucirumab | Part C: 200 mg Abemaciclib + 10mg/kg Ramucirumab Day1 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 or 150 or 200 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
Number analyzed (Participants) | 8 | 15 | 3 | 20 | 20 | 19 | 3 | 27 | 6 | 3 | 17
nanogram*hour/mL (ng*h/mL)
  Day 1: number analyzed (Participants) | 8 | 15 | 3 | 20 | 20 | 19 | 3 | 27 | 6 | 1 | 17
  Day 1 | 533 (69.6) | 979 (77.5) | 393 (31.0) | 886 (53.4) | 797 (69.0) | 1030 (127) | 394 (71.7) | 719 (77.3) | 967 (139) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of AUC = 482 ng*h/mL. | 518 (21.6)
  Steady State: number analyzed (Participants) | 1 | 8 | 1 | 3 | 11 | 6 | 2 | 10 | 0 | 0 | 10
  Steady State | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of AUC = 1350 ng*h/mL. | 3710 (41.1) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual value of AUC = 2270 ng*h/mL. | 2690 (53.4) | 1720 (119) | 1840 (115) | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of AUC = 1030 ng*h/mL and 1050 ng*h/mL. | 1550 (83.7) |  |  | 1400 (184)

11. Secondary Outcome: PK: Area Under the Concentration Curve (AUC) of Pemetrexed at Steady State in Part A
Description: Area under the plasma concentration versus time curve from time zero to infinity (AUC[0-∞]) of Pemetrexed in Part A was evaluated.
Time Frame: C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*hr/mL)
Arm/Group | Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed
Number analyzed (Participants) | 7 | 12
microgram*hour per milliliter (μg*hr/mL) | 201 (30) | 198 (32)

12. Secondary Outcome: PK: Area Under the Concentration Curve (AUC) of Active Gemcitabine Metabolite: 2',2'-Difluorodeoxyuridine (dFdU) on Day 1 and at Steady State (Cycle 2 Day 1) in Part B
Description: Area under the plasma concentration time curve from time zero to 12 hours (AUC[0-12h]) of active gemcitabine metabolite (dFdU) in Part B was evaluated
Time Frame: C1D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose; C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL (ng*h/mL)
Groups:
- 200 mg or MTD Abemaciclib + 1250 mg/m^2 Gemcitabine: 200 mg abemaciclib or maximum tolerated dose (MTD) under the combination treatment abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 mg/m^2 gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part B: 150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | 200 mg or MTD Abemaciclib + 1250 mg/m^2 Gemcitabine
Number analyzed (Participants) | 3 | 4 | 16
nanogram*hour/mL (ng*h/mL)
  Day 1: number analyzed (Participants) | 3 | 4 | 15
  Day 1 | 175000 (16) | 246000 (29) | 198000 (26)
  Steady State: number analyzed (Participants) | 2 | 3 | 8
  Steady State | NA (NA) — NA = Data reported as individual values when participants analyzed (n) were less than 3. Individual values of AUC[0-12h] = 201000 ng*h/mL and 249000 ng*h/mL. | 208000 (20) | 210000 (23)

13. Secondary Outcome: PK: Area Under the Concentration Curve (AUC) of LY3023414 in Part D
Description: Area under the plasma concentration versus time curve from time zero to infinity (AUC) of LY3023414 in Part D was evaluated. For Day 1, AUC is defined as AUC from time zero to infinity (AUC[0-∞]), for steady state, AUC is defined as AUC from time zero to the end of the dosing interval, tau (AUC[0-tau ])
Time Frame: C1D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose; C2D1 pre-dose and 1, 2, 4, 6, 8, 10 h post-dose
Population: All randomized participants who received at least one dose of study drug with evaluable PK data in Part D.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/mL (ng*h/mL)
Groups:
- Part D: 150 or 200 mg Abemaciclib + 150 mg LY3023414: 150 or 200 mg Abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 100 mg or 150 mg or 150 mg LY3023414 given orally every 12 hours on Days 1 through 21 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part D: 100 or 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 or 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414
Number analyzed (Participants) | 12 | 15 | 8
nanogram*hour/mL (ng*h/mL)
  Day 1 | 1005 (63) | 1751 (56) | 3809 (95)
  Steady State: number analyzed (Participants) | 12 | 4 | 1
  Steady State | 1303 (64) | 1293 (49) | NA (NA) — NA = No participants had sufficient PK data to compute AUC0-tau.

ADVERSE EVENTS:
Time Frame: Up to 4 years and 1 Month
Description: All randomized participants who received at least one dose of study drug in Part A, B, C, D and E. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 500 mg/m^2 pemetrexed given IV over approximately 10 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part B:150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 1250 mg/m^2 gemcitabine given intravenously over approximately 30 minutes on Days 1 and 8 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Day1: 150 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 mg/kg ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
- Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day1: 200 mg abemaciclib given orally every 12 hours on Days 1 through 21 of a 21-day cycle in combination with 10 mg/kg ramucirumab given intravenously over approximately 60 minutes on Day 1 of a 21-day cycle. Participants may continue to receive treatment until discontinuation criteria are met.
Arm/Group | Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed | Part B:150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Day1 | Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day1 | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 | Part D: 100 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 100 mg LY3023414 | Part D: 150 mg Abemaciclib + 150 mg LY3023414 | Part D: 200 mg Abemaciclib + 150 mg LY3023414 | Part D: 150 mg Abemaciclib + 200 mg LY3023414 | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 2/8 | 1/15 | 1/3 | 6/21 | 2/4 | 4/19 | 1/12 | 1/4 | 0/3 | 1/9 | 0/10 | 1/6 | 1/8 | 0/3 | 2/17
Serious Adverse Events (participants affected / at risk) | 4/8 | 8/15 | 1/3 | 10/21 | 3/4 | 12/19 | 3/12 | 3/4 | 1/3 | 2/9 | 3/10 | 0/6 | 4/8 | 0/3 | 9/17
Other Adverse Events (participants affected / at risk) | 8/8 | 15/15 | 3/3 | 21/21 | 4/4 | 19/19 | 12/12 | 4/4 | 3/3 | 8/9 | 10/10 | 5/6 | 8/8 | 3/3 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed (N=8) | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed (N=15) | Part B:150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine (N=3) | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine (N=21) | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Day1 (N=4) | Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day1 (N=19) | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 (N=12) | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 (N=4) | Part D: 100 mg Abemaciclib + 100 mg LY3023414 (N=3) | Part D: 150 mg Abemaciclib + 100 mg LY3023414 (N=9) | Part D: 150 mg Abemaciclib + 150 mg LY3023414 (N=10) | Part D: 200 mg Abemaciclib + 150 mg LY3023414 (N=6) | Part D: 150 mg Abemaciclib + 200 mg LY3023414 (N=8) | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab (N=3) | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 0/4 (0) | 0/10 (0) | 0 (0) | 1/10 (1) | 0/2 (0) | 0/9 (0) | 0/8 (0) | 0 (0) | 0/2 (0) | 0/4 (0) | 0/7 (0) | 0/4 (0) | 0/5 (0) | 0/2 (0) | 0/7 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial strain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A:150 mg Abemaciclib + 500 mg/m^2 Pemetrexed (N=8) | Part A: 200 mg Abemaciclib + 500 mg/m^2 Pemetrexed (N=15) | Part B:150 mg Abemaciclib + 1250 mg/m^2 Gemcitabine (N=3) | Part B: 200 mg Abemaciclib + 1250 mg/m^2 Gemcitabine (N=21) | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Day1 (N=4) | Part C: 200 mg Abemaciclib + 10 mg/kg Ramucirumab Day1 (N=19) | Part C: 150 mg Abemaciclib + 8 mg/kg Ramucirumab Days 1 and 8 (N=12) | Part C: 150 mg Abemaciclib + 10 mg/kg Ramucirumab Days 1 and 8 (N=4) | Part D: 100 mg Abemaciclib + 100 mg LY3023414 (N=3) | Part D: 150 mg Abemaciclib + 100 mg LY3023414 (N=9) | Part D: 150 mg Abemaciclib + 150 mg LY3023414 (N=10) | Part D: 200 mg Abemaciclib + 150 mg LY3023414 (N=6) | Part D: 150 mg Abemaciclib + 200 mg LY3023414 (N=8) | Part E: 100 mg Abemaciclib + 200 mg Pembrolizumab (N=3) | Part E: 150 mg Abemaciclib + 200 mg Pembrolizumab (N=17)
Anaemia (Blood and lymphatic system disorders) | 6 (20) | 12 (24) | 1 (2) | 10 (44) | 0 (0) | 5 (13) | 2 (3) | 0 (0) | 2 (3) | 3 (8) | 2 (2) | 0 (0) | 3 (3) | 2 (4) | 6 (12)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (10) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (6) | 4 (12) | 0 (0) | 3 (4) | 0 (0) | 3 (14) | 1 (14) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (5) | 0 (0) | 2 (2) | 1 (2) | 2 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (19) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (7) | 14 (31) | 1 (1) | 13 (28) | 2 (2) | 14 (32) | 10 (27) | 2 (3) | 2 (4) | 6 (6) | 9 (17) | 1 (1) | 6 (8) | 1 (1) | 10 (30)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (13) | 3 (3) | 13 (17) | 1 (2) | 12 (22) | 6 (11) | 2 (3) | 2 (2) | 5 (5) | 6 (16) | 3 (6) | 4 (6) | 0 (0) | 7 (7)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (18) | 0 (0) | 8 (10) | 1 (2) | 11 (17) | 3 (3) | 1 (2) | 2 (3) | 4 (5) | 7 (7) | 2 (4) | 6 (6) | 0 (0) | 4 (4)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (12) | 3 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (6)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (14) | 12 (32) | 2 (4) | 17 (30) | 2 (2) | 12 (23) | 5 (9) | 0 (0) | 2 (2) | 4 (7) | 4 (5) | 2 (2) | 2 (2) | 3 (4) | 12 (20)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Oedema peripheral (General disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 4 (8) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0/4 (0) | 0/10 (0) | 0 (0) | 1/10 (1) | 0/2 (0) | 0/9 (0) | 0/8 (0) | 0 (0) | 0/2 (0) | 0/4 (0) | 0/7 (0) | 0/4 (0) | 0/5 (0) | 0/2 (0) | 0/7 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 5 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural anxiety (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (4) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (13) | 3 (5) | 1 (2) | 4 (13) | 0 (0) | 4 (10) | 3 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (9) | 4 (17) | 2 (9) | 9 (36) | 0 (0) | 3 (7) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 3 (9) | 4 (7) | 1 (1) | 10 (24) | 0 (0) | 5 (13) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (3) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 3 (9) | 1 (3) | 0 (0) | 4 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 9 (17) | 0 (0) | 9 (12) | 1 (2) | 6 (7) | 6 (19) | 3 (8) | 1 (2) | 2 (2) | 3 (5) | 2 (2) | 5 (5) | 1 (1) | 9 (20)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (6) | 1 (2) | 7 (8) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid intake reduced (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 0 (0) | 4 (6) | 0 (0) | 1 (2) | 1 (8) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (12)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (4) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (5) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (3) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial spasm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological decompensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0/4 (0) | 0/5 (0) | 0/0 (0) | 0/11 (0) | 0/2 (0) | 0/10 (0) | 1/4 (1) | 0/0 (0) | 0/1 (0) | 0/5 (0) | 0/3 (0) | 0/2 (0) | 0/3 (0) | 0/1 (0) | 0/10 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (8) | 1 (1) | 5 (9) | 0 (0) | 5 (5) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (10) | 1 (1) | 3 (3) | 1 (2) | 2 (4) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 3 (5) | 0 (0) | 4 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (15) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (10) | 0 (0) | 1 (3) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02079636/SAP_000.pdf
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT02079636/Prot_001.pdf